CLINICAL TRIAL: NCT01383525
Title: Direct Application of Selective Laser Trabeculoplasty in Open Angle Glaucoma . Single Site Study
Brief Title: Direct Application of Selective Laser Trabeculoplasty in Open Angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BelkinVision (Industry)
Collaborators: Horizon 2020 - European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-11-8414
Record Dates: First submitted 2011-06-22; First posted 2011-06-28 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Glaucoma
Keywords: SLT, LTP, DSLT; non contact; Trabeculoplasty; Laser; intraocular pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Masking Description: No masking for treatment. The follow-up and primary endpoint assessment, intra-ocular pressure (IOP) measurement, is performed by masked ophthalmologist.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Direct Selective Trabeculoplasty (Experimental): Treatment by an Direct Selective Trabeculoplasty device
  Interventions: Device: Direct Selective Trabeculoplasty device

INTERVENTIONS:
Device: Direct Selective Trabeculoplasty device — Patients will be treated with a Direct Selective Trabeculoplasty (DLTP) laser. Placement of the spots is on the sclera around the limbus.

SUMMARY:
The trial objectives are to establish the safety & efficacy of using a DLTP laser to perform laser trabeculoplasty to reduce Intraocular Pressure (IOP) in patients with open angle glaucoma (Including Pigmentary & Exfoliative Glaucoma), that did not achieve adequate IOP control by conventional therapy.

DETAILED DESCRIPTION:
This is a single site outpatient feasibility study assessing the safety & efficacy of the DLTP laser in the ability to reduce IOP in patients with open angle glaucoma (OAG). The investigational site will accrue patients with uncontrolled OAG. These eyes will be treated with the direct application of Direct Laser Trabeculoplasty (DLTP)/ Direct Selective Laser Trabeculoplasty automated device (DSLT).

Only one eye per patient is to be treated with the investigational device during the study.

The laser parameters used will be like these used in the Selective trabeculoplasty (SLT) device (CE/FDA approved), but all laser beams will be applied in about one-second, through the peri-limbal.

Subjects will be evaluated preoperatively and postoperatively at 1 hour, 2 hours (and hourly to 4 hours in the event of an IOP elevation in the immediate postop course), 1 day, 1 week, and 1, 3, 6 months.

Patients will be followed out to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient is aged 18 years or older, with 2 sighted eyes.
* Eye to be treated have average IOP *22 mmHg, measured at 2 pretreatment visits.
* Eye to be treated either exhibits:
* poorly controlled open angle glaucoma including Pigmentary & Exfoliative Glaucoma
* Patient would be considered eligible for conventional laser trabeculoplasty.
* Patient is willing to participate in the 6-month study and to adhere to the follow-up schedule.
* Patient is willing to review and sign a consent form.

Exclusion Criteria:

* evidence of glaucoma other than open-angle glaucoma;
* severe para-central or generalized field defect;
* Any ocular condition that precluded adequate visualization and treatment of the trabecular meshwork.
* Prior glaucoma surgery other than laser trabeculoplasty or peripheral iridotomy.
* Patient has mental impairment such that he/she could not understand the protocol or is not in a position to provide written informed consent.
* Patient is pregnant.
* Patient might require other ocular surgery within the 6-month follow-up period.
* Patient has a medical history that suggested the potential for complications from Direct Selective Trabeculoplasty (DSLT)
* Having concurrent treatment with systemic steroids.
* Patient is under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-07; Primary Completion 2019-08 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Reduction of Intra-Ocular pressure | 1,3 month
  Percentage reduction of intra-ocular pressure following the non contact selective laser trabeculoplasty treatment

SECONDARY OUTCOMES:
Reduction of Intra-Ocular pressure | 6 months
  Percentage reduction of intra-ocular pressure following the non contact selective laser trabeculoplasty treatment

OTHER OUTCOMES:
Number of medications | 6 months
  Number of medications after treatment, as compared to before treatment.
Physician perception of the usability of the system. | 1 month
  Physician perception of the usability of the system.

CONTACTS AND LOCATIONS:
Overall Officials: Alon Skaat, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- The Sam Rothberg Glaucoma Center Goldschleger Eye Institute Sheba meical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No